CLINICAL TRIAL: NCT03873298
Title: The Influence of Inhaled Nitric Oxide on Oxygen Saturation of Patients With COPD and IPF During Six Minute Walk Test.
Brief Title: Inhaled NO in IPF and COPD During 6 Minute Walk Test
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Collaborators: Bellerophon (Industry)
Responsible Party: Principal Investigator, Mordechai Kremer, Head of the pulmonary division, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0135-18-rmc
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: COPD; IPF; Inhaled Nitric Oxide; Six Minute Walk Test; Oxygen Saturation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: RCT, placebo controlled
Who Masked: Participant
Masking Description: The participants don't know if the cartridge used in the INO device is placebo or NO
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- COPD (Experimental): Each participant will undergo two six minute walk tests and the results will be compared within each subject.
  Interventions: Drug: Inhaled nitric oxide
- IPF (Experimental): Each participant will undergo two six minute walk tests and the results will be compared within each subject.
  Interventions: Drug: Inhaled nitric oxide

INTERVENTIONS:
Drug: Inhaled nitric oxide — Inhaled nitric oxide delivered through a pulsatile nitric oxide drug delivery system

SUMMARY:
Our objective is to evaluate the influence of inhaled NO on the saturation and exercise capacity of patients with COPD and IPF. each participant will undergo two six minute walk tests, one with inhaled NO and the other with placebo.

DETAILED DESCRIPTION:
This is a randomiized, placebo controlled trail that will evaluate the influence of inhaled NO (INO) on the saturation and exercise capacity of patients with COPD and IPF. All patients will sign a consent form before enrolment. Each patient will undergo two six-minute walk tests. Whether the INO will be used in the first or the second trial will be determined by computer generated randomization with random numbers sealed in opaque envelops. For the placebo 6-minute test we will use placebo cartridges in the INO generator, for INO 6-minute test we will use NO cartridges. The treatment with INO or placebo will start 20 minutes before the 6-minute walk test and will end at the end of the 6-minute walk test. Between tests a time interval of at least 60 minutes will be kept. During the test, the patients' pulse and saturation level will be monitored with a pulse oximetry. The data will be recorded continuously from baseline to 5 minutes after the test is over. The distance the patient walked will also be recorded. Patients that require supplemental oxygen will perform the tests with oxygen supplementation.

Dosing The NO dosing will be fixed. The first 10 patients will be treated with INO at a dose of 45 parts per million (ppm) per kilogram (kg). from patient 10 to 20 a dose of 75 ppm per kg will be given and from patient 20-100 a dose of 115 ppm per kg will be given.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with COPD with disease severity of GOLD stage 3-4
2. Patients with IPF with a Forced vital capacity under 80% and a diffusion capacity under 60%
3. Ambulatory patients that can perform a 6-minute walk test

Exclusion Criteria:

1. Patients with moderate to severe heart failure - EF < 40%
2. Patients with severe PVD or scleroderma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-03-04 (Actual); Primary Completion 2020-03-04 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Saturation level during the test | 26 minutes
  AUC of the saturation value during six minute walk test

CONTACTS AND LOCATIONS:
Overall Officials: Mordechai Kramer, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Freidkin L, Kramer MR, Rosengarten D, Izhakian S, Taieb S, Pertzov B. The acute effect of inhaled nitric oxide on the exercise capacity of patients with advanced interstitial lung disease: a randomized controlled trial. BMC Pulm Med. 2024 May 10;24(1):226. doi: 10.1186/s12890-024-03051-4. PMID 38724947